CLINICAL TRIAL: NCT05895318
Title: Perceptions of MDMA-Assisted Therapy Among Veterans With PTSD
Acronym: PMATAVP
Status: Completed | Type: Observational
Sponsor: Albany Research Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 061006
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: MDMA; MDMA-Assisted Therapy; Psychedelic; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this exploratory, mixed-method design study is to gather qualitative and quantitative data obtained through interviews and questionnaires with veterans who are currently enrolled at the VA for healthcare. The main question this study aims to answer is: How do veterans diagnosed with PTSD and enrolled for care at the VA understand MDMA-assisted therapy for PTSD? Using a story-completion approach, participants will be provided with a brief story starter involving a fictitious character and scenario and asking them to complete the story. Few contextual details will be offered about the character. In responding to ambiguous cues, participants are thought to project their conscious and subconscious perceptions about the phenomenon in question onto the story, a useful method for exploring stigmatized topics. The purpose of this exercise is to ascertain the participants attitudes and perceptions regarding MDMA-Assisted Therapy.

DETAILED DESCRIPTION:
Veterans will be informed of the study by their VA providers (Behavioral Health Clinic, PCMHI, PTSD Clinic, CDRP, Primary Care). Veterans who are interested will have their contact information passed on to the study investigators. Once screened and enrolled in the study veterans will complete a brief demographics form, and three brief symptom screening questionnaires: PTSD Checklist for DSM-5, 5-Item screener for PTSD, and Patient Health Questionnaire 9. Participants then engage in the recorded interview during which they are provided with a brief story starter, as described above. In the story, a fictitious veteran with a diagnosis of PTSD is offered an opportunity to enroll in a clinical trial and receive MDMA-Assisted therapy. Participants are asked to share what questions, concerns, hopes, and expectations may be present for the fictitious veteran in the story. Interviews will then be transcribed and the PI and the collaborators will read all transcriptions and generate recurring themes that can be reliably coded. The investigators will then code the transcripts for the presence of themes. Data analytic plans include calculating the prevalence of each theme and examining their correlates with measures of severity of symptoms as well as any demographic variables. It is hoped that this data can inform educational and other roll-out efforts within the VA system as MDMA-Assisted therapy approaches FDA approval as a treatment for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in VA care
* Active diagnosis of PTSD, as determined by the referring provider or confirmed by medical records.
* Age 18 or older
* Fluent in written and spoken English

Exclusion Criteria:

* Cognitively impaired to the extent that patient cannot comprehend the survey
* Has already completed the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The demographic makeup of the sample mimics the demographic makeup of the population of veterans served by VA. As such, the racial distributions will likely be primarily Caucasian, the sample is likely to be predominantly male, ranging in age from 20-100, with an average of 58 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 | 2 weeks
  Screening tool for depressive symptoms. Scores range from 0-27 with lower scores indicating better outcomes
PTSD Checklist for DSM5 | 4 weeks
  Screening tool for PTSD symptoms. Scores range from 0-80 with lower scores indicating better outcomes
5 Item Screener for PTSD | 2 weeks
  Screening tool for PTSD symptoms. Scores range from 0-4 with lower scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Holley, Ph.D., Principal Investigator — Stratton VA Medical Center
Locations (1):
- Stratton VA Medical Center, Albany, New York, United States